CLINICAL TRIAL: NCT00719407
Title: Neonatal Erythropoietin in Asphyxiated Term Newborns: a Phase I Trial
Brief Title: Neonatal Erythropoietin in Asphyxiated Term Newborns
Acronym: NEAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Thrasher Research Fund (Other); UCSF Benioff Children's Hospital Oakland (Other); University of Washington (Other); Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Principal Investigator, Yvonne Wu, Professor of Neurology and Pediatrics, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H9299-32566-01; Thrasher 02827-0
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Hypoxic-ischemic Encephalopathy
Keywords: birth asphyxia; neonatal encephalopathy; hypoxic-ischemic encephalopathy; neuroprotection; neonate
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum | interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All enrolled patients will be in this single arm, who will receive experimental drug treatment.
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — 250 U/kg/dose x 6 doses (n=3); 500 U/kg/dose x 6 doses (n=6); 1,000 U/kg/dose x 6 doses (n=7) 2,500 U/kg/dose x 6 doses (n=8)
  Other Names: Procrit

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of moderate to high doses of erythropoietin in newborn infants with birth asphyxia.

DETAILED DESCRIPTION:
Newborn infants with birth asphyxia are at high risk of death or long-term neurologic disability; yet therapies for birth asphyxia are currently limited. Erythropoietin (Epo) is a FDA-approved drug that is an effective neuroprotective agent in animal models of birth asphyxia. This is a phase I dose finding multi-center trial that will test the safety and pharmacokinetics of Epo in human infants with birth asphyxia. The long-term objectives of the proposed research are to reduce mortality and to decrease the risk of long-term disabilities in infants who survive beyond the newborn period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 36 weeks gestational age
2. Perinatal depression (low Apgar score, need for resuscitation)
3. Moderate to severe encephalopathy

Exclusion Criteria:

1. Specific aEEG findings
2. Intrauterine growth restriction
3. Severe congenital anomaly, genetic syndrome, metabolic disorder, arthrogryposis, TORCH infection
4. Microcephaly
5. Infant older than 23.5 hours of age at the time of consent
6. Infant judged by an attending physician to be likely to die due to the severity of illness
7. Polycythemia
8. Hypertension
9. No in-dwelling line

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Serious adverse event | 14 days of life

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 1 to 11 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne W Wu, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Rogers EE, Bonifacio SL, Glass HC, Juul SE, Chang T, Mayock DE, Durand DJ, Song D, Barkovich AJ, Ballard RA, Wu YW. Erythropoietin and hypothermia for hypoxic-ischemic encephalopathy. Pediatr Neurol. 2014 Nov;51(5):657-62. doi: 10.1016/j.pediatrneurol.2014.08.010. Epub 2014 Aug 27. PMID 25439577
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452
- [Derived] Wu YW, Bauer LA, Ballard RA, Ferriero DM, Glidden DV, Mayock DE, Chang T, Durand DJ, Song D, Bonifacio SL, Gonzalez FF, Glass HC, Juul SE. Erythropoietin for neuroprotection in neonatal encephalopathy: safety and pharmacokinetics. Pediatrics. 2012 Oct;130(4):683-91. doi: 10.1542/peds.2012-0498. Epub 2012 Sep 24. PMID 23008465